CLINICAL TRIAL: NCT00624611
Title: Post Cardiac Surgery Blood Loss: Effect of Washing Residual Cardiopulmonary Bypass Circuit Blood Red Cells Prior to Re-infusion. A Proof of Concept Study
Brief Title: The Effect of Washing Red Blood Cells on Post Heart Surgery Blood Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Norbert Froese, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H07-01444
Record Dates: First submitted 2008-02-13; First posted 2008-02-27 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Cardiopulmonary Bypass
Keywords: CPB; red blood cell washing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Residual pump blood management post aortic cannula removal
  Interventions: Procedure: Residual pump blood management post aortic cannula removal
- 2 (Experimental): Residual pump blood management post aortic cannula removal
  Interventions: Procedure: Residual pump blood management post aortic cannula removal

INTERVENTIONS:
Procedure: Residual pump blood management post aortic cannula removal — Residual pump blood will be maximally hemoconcentrated by further ultrafiltation within the CPB machine. Resulting hematocrit will be approximately 0.4. The total residual pump blood volume, approximately 300ml, will be reinfused over one hour, beginning 15 minutes after removal of the aortic cross clamp. Additional protamine sulfate will be given every 30 minutes during the infusion, .03 mg/ml of residual pump blood. Procedures in this group do not deviate from current standard practice.
  Arms: 1
Procedure: Residual pump blood management post aortic cannula removal — All residual pump blood will be processed with a bedside red cell washing device (Cell Saver). The resulting total volume of concentrated red cells will be infused over one hour, beginning 15 minutes after removal of the aortic cross clamp. Administration of additional protamine is not required due to the low concentrations of heparin in the resulting product.
  Arms: 2

SUMMARY:
When a child undergoes heart surgery, a heart lung machine is used to keep blood flowing while the child's own heart is stopped. After surgery, a significant amount of the child's own blood is left in this machine. In the case of small children, the relative amount of blood potentially lost to the child in this way is very large.

In older children, and those who have undergone less complicated surgery, this blood can all returned to the child. Giving the child back his or her own blood makes is less likely that the child will need a transfusion of donated blood.

However, in younger children, or in children who have undergone more complicated surgery, most or all of this blood is thrown away. This is because of worry that returning this blood may cause bleeding, and excessive bleeding is one of the most feared complications of heart surgery.

This project will explore a method whereby the red blood cells left in the heart lung machine can be returned to children without increasing the risk of bleeding. It will also carefully examine the exact causes of higher bleeding risk in children getting their own blood back so that in the future, all children can have their own blood returned at the end of surgery.

DETAILED DESCRIPTION:
The primary hypothesis of this study is that in our study population, compared to re-infusion of residual CPB blood, re-infusion of only the red cell component of residual CPB blood, causes a lesser defect in clotting, leading to decreased hemorrhage and less post-operative blood loss.

The secondary objectives of this project are to document the effects on the clotting system of pump blood re-infusion by means of in laboratory testing. This work has not been done and is of crucial importance to future optimization of the use of pump blood. We expect to detect and quantify with significant accuracy any increased bleeding risk with our hemostatic profiling. This information will be invaluable in planning the safe introduction of residual CPB blood re-infusion smaller children and those with increase risk of postoperative blood loss. Furthermore, we will determine whether or not any of the potentially beneficial effects to the clotting system of returning all components of residual CPB blood, such as an increase in functioning platelets, or an increase in clotting factors, are realized. This information will determine the utility of pursuing means by which these non red cell components of residual CPB blood can be safely re-infused.

Induction of anesthesia, arterial and venous vascular catheter placement, heparin administration, cardiopulmonary bypass machine setup and priming, conduct of CPB, ultrafiltration of blood during CPB, post-CPB protamine administration and post-CPB blood ultrafiltration will all be standardized as per current clinical practice.

Residual CPB blood will be processed and re-infused according to group allocation.

Intravascular volume in the form of crystalloid, and blood products will be administered over and above the study residual blood product infusion as required according to protocol.

Subjects will have blood sampled for hemoglobin concentration immediately after induction of anesthesia and again 24 hours following their surgery.

Arterial blood will be sampled from the patient for a hemostatic profile, outlined in the adjacent text box, after separation from CPB and prior to initiation of residual CPB blood product re-infusion. A second sample will be obtained when re-infusion of residual CPB blood product is complete. In addition, a hemostatic profile will be run directly on a sample of the residual CPB blood product.

Subject demographic data, surgical diagnosis and procedures, CPB data, all medication, blood product and intravenous fluid administration, total volume of study fluid administered, blood lost during surgery to sponges and suction and 24 hour mediastinal drainage will be recorded for all subjects. Any cases of incomplete re-infusion of study blood product will be noted as will the reason for the occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Children between 15 and 30 kg undergoing cardiac surgery requiring cardiopulmonary bypass at British Columbia's Children's Hospital.
* All children will be between 2 and 10 years of age.
* Surgery will only involve single atriotomy.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Total perioperative blood loss | During surgery

SECONDARY OUTCOMES:
Components of the hemostatic profile will be compared between groups as secondary outcome variables | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Froese, MD, Principal Investigator — University of British Columbia; John Wu, Study Director — University of British Columbia; Jacques LeBlanc, Study Director — University of British Columbia; Andrew Campbell, Study Director — University of British Columbia; Doug Salt, Study Director — University of British Columbia; Pascal Lavoie, Study Director — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada